CLINICAL TRIAL: NCT01864642
Title: A Study of the Effects of a Single Osteopathic Manipulative Treatment (OMT) on Intraocular Pressure (IOP)in Un-medicated Confirmed Ocular Hypertensive (OHT) or Glaucoma Suspect Subjects
Brief Title: Effects of a Single OMT on Intraocular Pressure (IOP) in Ocular Hypertenive or Glaucoma Suspect Subjects
Acronym: OMT4OHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UW IRB 2012-1102
Record Dates: First submitted 2013-05-20; First posted 2013-05-29 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- osteopathic manipulative treatment (Experimental): osteopathic manipulative treatment (OMT)
  Interventions: Procedure: osteopathic manipulative treatment (OMT)

INTERVENTIONS:
Procedure: osteopathic manipulative treatment (OMT)
Procedure: osteopathic manipulative treatment (OMT) — OMT is a form of manual medicine performed by osteopathic physicians
  Other Names: OMT is a form of manual medicine

SUMMARY:
The hypothesis is that osteopathic manipulative treatment (OMT)will significantly reduce intraocular pressure (IOP) in individuals with ocular hypertension (OHT) and glaucoma suspect patients.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of irreversible blindness in the United States and the world. Approximately 2.8 million Americans have been diagnosed with glaucoma. Based on pilot studies and the clinical experience of the PI, a power analysis indicated that in order to lower IOP by 4 mm Hg 28 subjects would be needed, 14 in the experimental group and 14 in the control/comparator group.

The intervention is OMT. Based on the anatomy of the eye and the dysfunctions underlying primary open angle glaucoma (POAG), the presumed mechanisms are one or the other or a combination of the following. 1) Anatomic: the OMT benefit may occur by the biomechanical restoration of drainage through the trabecular meshwork and Schlemm's canal. 2) Neurologic: the OMT may affect the parasympathetic innervations from the Edinger-Westphal fibers via the cranial nerve III as well as the sympathetic innervations arising in the T1 to T3 levels then via the superior cervical ganglion which then course to the eye.

The OMT protocol takes 25-27 minutes to administer and addresses cranial, cervical, upper body, spinal and sacral structures designed to affect the anatomic, physiologic processes (e.g. lymphatic drainage from the neck and face), neurologic structures (sympathic and parasympathetic) affecting visual processes. A very similar OMT protocol was used in a study on healthy elder and resulted in improved balance and equilibrium. In that study there were no adverse outcomes reported.

The control/comparator subjects will lay on the OMT table for the same 25-27 minutes in the same time periods in which experimental subjects were in the prone, lateral recumbent, and supine positions.

ELIGIBILITY:
Inclusion Criteria:

Subject inclusion criteria.

1. Subjects will be of either sex, age 18 years or older, and of any race or eye color.
2. Subjects with confirmed ocular hypertension (OHT) or glaucoma suspects whose IOP was ≥ 20 mmHg at two measurements separated by at least 3 months.
3. Subjects who do not have visual field defect(s), as determined by Visual Field Analysis within the last year.
4. Subjects who do not have abnormal cupping of the optic nerve head.
5. Subjects who do not have narrow angles as determined by gonioscopy (must be at least angle grade 2 to 3; Shaffer Classification Scale) recorded in the subject's patient record or as determined by biomicroscopy.
6. Subjects who have not been treated with ocular hypotensive agents (or, if they have been treated, not for at least the preceding 3 months). In essence, the subjects will have been and be undergoing "watchful waiting" by their eye care practitioner(s) because no definitive diagnosis of glaucoma requiring treatment has been made.
7. Subjects must satisfy all informed consent requirements. 8 Subjects whose mean IOP measurements in at least one (1) eye, the same eye(s), must be:

9. Greater than or equal to 20 mmHg at the 8 AM time-point on the Screening and Enrollment Visits (1 and 2) and 10. Greater than or equal to 19 mmHg at the 10 AM, 12 Noon, and 4 PM time-points on the Screening and Enrollment Visits (1 and 2).

-

Exclusion Criteria:

1. Subjects who have had any traumatic brain injury or head trauma, which resulted in upper-spinal fusion and/or cranial bone surgery, which implanted a metal plate.
2. Subjects who have a concurrent diagnosis of cancer or metastatic disease affecting the head and neck.
3. Subjects who have been diagnosed with glaucoma or ocular hypertension and whose condition requires medical treatment other than "watchful waiting."
4. Subjects who are less than 18 years old.
5. Subjects who are lactating, pregnant, or plan to become pregnant in the time planned for the study.
6. Subjects who have a history of chronic or recurrent severe inflammatory eye disease (e.g., scleritis, uveitis) in either eye as determined by patient history and/or examination.
7. Subjects who have a history of clinically significant or progressive retinal disease in either eye such as retinal degeneration, diabetic retinopathy, or retinal detachment with permanent field loss as determined by patient history and/or examination.
8. Subjects who have a history of serious ocular trauma in either eye within the past six (6) months as determined by patient history and/or examination.
9. Subjects who have had intraocular surgery in either eye within the past six (6) months as determined by patient history and/or examination.
10. Subjects who have had ocular laser surgery in either eye within the past three (3) months as determined by patient history and/or examination.
11. Subjects who have a history of ocular infection or ocular inflammation in either eye within the past three (3) months as determined by patient history and/or examination.
12. Subjects who have any abnormality preventing reliable applanation tonometry of either eye (e.g., keratoconus, corneal or conjunctival scarring).
13. Subjects who have any abnormality preventing reliable assessment of pupil diameter in either eye (e.g., congenital pupil anomaly, posterior synechiae, anterior cleavage syndrome, afferent defects, prior surgery, etc.).
14. Subjects who have less than a thirty (30) days stable dosing regimen before the Screening and Enrollment Visits (Visits 1 and 2) of any non-ocular medications that may affect IOP, administered by any route and used on a chronic basis. These may include, but are not limited to, alpha agonists, beta-blockers, calcium channel blockers, antimuscarinic agents, and phenothiazines.
15. Subjects who have other treatments and/or surgeries unrelated to the eye condition scheduled in the time planned for the study.
16. Subjects who are allergic to Latex, PABA, Proparacaine, or Fluorescein.
17. Subjects who have had prior surgical or laser treatment for the purpose of lowering their IOP.
18. Subjects who currently have systemic infections resulting in fever or immunosuppression.
19. Subjects who have had previous OMT, chiropractic manipulation, massage, or other forms of manual therapy within the last 2 months.
20. Subjects who are unable to give appropriate informed consent due to mental or other limitations.
21. Additionally, the Principal Investigator may declare any subject ineligible for a valid medical reason.

    -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | up to 3 days
  Goldman Tonometry

SECONDARY OUTCOMES:
pupillometry | measured on day one and two to assess eligibility, assess on day three at the time of the intervention, then on day 7 as last day of subject participation (up to 7 days)
  Pupillometry measures the pupil size and reactivity to light

CONTACTS AND LOCATIONS:
Overall Officials: Hollis H King, DO, PhD, Principal Investigator — Univ Wisconsin Dept of Family Medicine
Locations (1):
- UW Dept of Ophthalmology Clinic, Madison, Wisconsin, United States